CLINICAL TRIAL: NCT06292767
Title: The Impact of Two Different Mechanical Ventilation Strategies During Cardiopulmonary Bypass on Mechanical Power and Postoperative Pulmonary Complications
Brief Title: Cardiopulmonary Bypass on Mechanical Power and Postoperative Pulmonary Complications
Status: Completed | Type: Observational
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Gamze Talih, CLINICAL PROFESSOR, TC Erciyes University
Other Study IDs: 2023/462
Record Dates: First submitted 2024-01-24; First posted 2024-03-05 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Postoperative Pulmonary Atelectasis; Pneumothorax; Pneumonia; Ards; Respiratory Failure
MeSH Terms: conditions — Pulmonary Atelectasis; Pneumothorax; Pneumonia; Acute Lung Injury; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Not ventilated: Non-ventilated patient group.Patients will be placed in the cardiac bypass mode of the anesthesia machine. Only 150 ml of free air flow will be provided and mechanical ventilation will be turned off.
  Interventions: Other: mechanical power calculation
- Ventilated: Patients will continue to be ventilated at Fraction of inspired oxygen(FiO2): 40%, Tidal volume(TV): 3 ml/kg, frequency 12 breaths/min, Positive end expiratory pressure (Peep): 5 cm/H2O.
  Interventions: Other: mechanical power calculation

INTERVENTIONS:
Other: mechanical power calculation — Mechanical Power= 0.098×Minute ventilation× (peak pressure - 0.5 (plato pressure-PEEP)). These parameters are monitored on the monitor while the patient is mechanically ventilated and placed into the equation

SUMMARY:
During cardiopulmonary bypass (CPB), oxygenation of the patient on the pump can be left completely under pump control, or the lungs can be ventilated with low tidal volume to reduce atelectasis. In recent years, the concept of mechanical power has been used to determine the extent of ventilator-related lung damage. This concept of mechanical power, by which the energy transferred by the ventilator to the lungs can be calculated, will be measured at certain intervals in CPB surgery patients on the pump and compared between the two groups. The investigators aimed to investigate the effect of two different ventilation methods on mechanical power and its relationship with postoperative pulmonary complications.

DETAILED DESCRIPTION:
Patients will be taken to the operating table after preoperative evaluation. Routine monitoring and routine anesthesia method will be applied to the patient. Access will be made through the radial artery for arterial catheterization. Patients will be ventilated with 6-8 ml/kg tidal volume, 12-14 frequency/min, 5 Positive end expiratory pressure(PEEP), 60% Fraction of inspired oxygen(FiO2) and oxygen saturation over 94. End tidal Carbon dixide(CO2) will be kept in the range of 32-37. After cardiac catheterizations are performed, the pump will be entered, and after all preparations are completed, an aortic cross-clamp will be placed and cardioplegic solution will be sent. After the patient enters the pump at full flow; Group 1: Non-ventilated patient group. Here, patients will be placed in the cardiac bypass mode of the anesthesia machine. Only 150 ml of free air flow will be provided and mechanical ventilation will be turned off.

Group 2: Patients will continue to be ventilated at FiO2: 40%, TV: 3 ml/kg, frequency 12 breaths/min, peep: 5 cm/H2O.

ELIGIBILITY:
İnclusion criteria:

* Patients who will undergo elective cardiopulmonary bypass surgery and agree to participate in the study
* Patients who will undergo coronary or valve surgery
* Surgeries performed on a stopped heart
* Patients over 18 years

Exclusion criteria:

* Patients undergoing emergency cardiac surgery
* Patients who will undergo redo surgery
* Patients who will undergo total circulatory arrest surgery
* Patients in a state of preoperative shock
* Patients with acute and chronic hypoxemia (PaO2 <65mmHg, SpO2 <95 in room air)
* Patients followed with mechanical ventilation for 7 days before surgery
* Patients with BMI>35
* Patients with obstructive sleep apnea syndrome
* Patients with pulmonary artery pressure >50 mmHg
* Patients with glomerular filtration rate <30 ml/min

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are over 18 years and agree to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2024-03-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-04-25 (Actual)

PRIMARY OUTCOMES:
mechanical power | intraoperative
  mechanical power=0.098*minute ventilation *(Ppeak-0.5*(Pplato-PEEP)

SECONDARY OUTCOMES:
mechanical power | postoperative in intensive care unit
  mechanical power=0.098*minute ventilation *(Ppeak-0.5*(Pplato-PEEP)

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Kayseri, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No